CLINICAL TRIAL: NCT07369050
Title: Is the Provox ActiValve Only a Problem Solver? A Randomized Trial Comparing Routine Use of the ActiValve to Standard Voice Prostheses After Total Laryngectomy With Tracheoesophageal Puncture
Brief Title: A Randomized Trial Comparing Routine Use of the ActiValve to Standard Voice Prostheses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1610; NCI-2026-00404 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Routine "as needed" exchange with Provox ActiValve (Experimental): Participants randomized to Arm 1 will receive a Provox® ActiValve® at the first VP replacement after randomization
  Interventions: Device: Provox® ActiValve®
- Standard indwelling VP with optional cross-over to Provox ActiValve (Experimental): Participants randomized into Arm 2 will receive their standard VP exchanges on "as needed" basis through the 12-month study period.
  Interventions: Device: Provox® ActiValve®
- Prophylactic Provox ActiValve exchange (Experimental): Participants randomized to Arm 3 will receive a Provox® ActiValve® at the first VP replacement after randomization and prophylactic exchange will target replacement of the device between 9 months +/-1 month after fit.
  Interventions: Device: Provox® ActiValve®

INTERVENTIONS:
Device: Provox® ActiValve® — Participants experiencing early leakage with previous voice prostheses (device life less than 4-8 weeks). The device reduced the need for frequent replacements in a majority of users but not in all"7. The Light valve strength will be used in this trial.

SUMMARY:
The goal of this clinical research study is to learn if regular use of Provox® ActiValve® by patients after a total laryngectomy with TEP can decrease the number of VP device replacements needed annually.

DETAILED DESCRIPTION:
Primary Objective:

To determine whether routine use of Provox® ActiValve® voice prosthesis decreases annual number of clinical procedures to exchange VP in indwelling voice prosthesis users after total laryngectomy with TEP.

Secondary Objectives:

1. To compare outcomes, adverse events, and costs associated with routine use of Provox® ActiValve® (experimental) versus standard indwelling voice prostheses (comparator)
2. To compare outcomes, adverse events, and costs associated with prophylactic exchange of Provox® ActiValve® versus routine use of Provox® ActiValve® (experimental) or standard indwelling voice prostheses (comparator)

Exploratory objectives:

1. To explore relationships between clinicodemographic features and device/TEP function
2. To explore relationships between pharyngoesophageal pressures via manometry and device/TEP function
3. To explore relationships between oral/tracheal microbiome and device/TEP function
4. To describe novel use of prophylactic exchange of Provox® ActiValve®

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age status post total laryngectomy with tracheoesophageal puncture
2. Using or ready for fit of indwelling voice prosthesis
3. No evidence of disease (NED) in head and neck
4. At least 6 months since cancer treatment
5. TEP tract length 4.5 to 12.5mm at time of enrollment*

   * The range reflects the available device sizes for the Provox® ActiValve® . Eligibility is determined by confirming that the patient is appropriately fitted with a VP within this size range, based on the site's standard clinical practice (e.g. appearance/fit and/or depth gauge).

Exclusion Criteria:

1. History of recurrent leak around voice prosthesis and/or severely enlarged puncture (within last 12 months)
2. History of recurrent VP extrusion (within last 12 months)
3. Currently using specialty Activalve voice prosthesis as a "problem solver" due to poor device life as defined in the Instructions for Use (IFU)
4. History of recurrent early VP leak within 4 to 8 weeks of fit (within last 12 months)
5. Active malignancy in head and neck and/or chest at the time of enrollment
6. Receiving or planned for head and neck radiation therapy (RT) at the time of enrollment
7. Receiving regular magnetic resonance imaging (MRI) for cancer surveillance or other medical reasons
8. Planned regular VP exchanges at outside facility within next 12 months
9. History of gastric pull-up reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Hutcheson, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org